

#### **Informed Consent**

# INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH WITH OPTIONAL PROCEDURES

A Pilot Trial of Pembrolizumab Plus Chemoradiotherapy in Participants with Unresectable Gastroesophageal Cancer 2019-1253

| Subtitle: MK3475-901 US Main ICF v9 | diskriggistatelististuummuutuum geestaatista aa aa taa aa |
|---|---|
| Study Chair: Jaffer A. Ajani | |
| Participant's Name | Medical Record Number |

This is an informed consent and authorization form for a research study. It includes a summary about the study. A more detailed description of procedures and risks is provided after the summary.

This research has been reviewed and approved by an Institutional Review Board (IRB - a committee that reviews research studies).

## STUDY SUMMARY

The goal of this clinical research study is to learn if pembrolizumab in combination with mFOLFOX6 (5-fluorouracil and oxaliplatin), docetaxel, and radiation therapy can help to control gastroesophageal cancer. The safety of this combination will also be studied.

**This is an investigational study.** Pembrolizumab is FDA approved and commercially available for the treatment of gastroesophageal cancer. Docetaxel, oxaliplatin, and 5-fluorouracil are FDA approved and commercially available for the treatment of gastroesophageal cancer. Radiation therapy is delivered using FDA approved and commercially approved methods.

The combination of pembrolizumab, mFOLFOX6, and radiation therapy is considered investigational. The study doctor can explain how the study drugs are designed to work.

The study drugs may help to control the disease. Future patients may benefit from what is learned. There may be no benefits for you in this study.

Your participation is completely voluntary. Before choosing to take part in this study, you should discuss with the study team any concerns you may have, including side effects, potential expenses, frequent visits to the clinic, and time commitment.

You can read a list of potential side effects below in the Possible Risks section of this consent.

You may receive pembrolizumab for up to 20 study cycles. You may receive mFOLFOX6 for up to 8 weeks. You may receive 5-FU, docetaxel, and radiation for up to 5 weeks.

Pembrolizumab will be provided at no cost to you while you are on study. You and/or your insurance provider will be responsible for the cost of mFOLFOX6, docetaxel, and radiation therapy.

You may choose not to take part in this study. Instead of taking part in the study, you may choose to receive 5-fluorouracil, docetaxel, or oxaliplatin outside of this study. The study doctor will discuss with you the risks and benefits of these treatments. You may choose to receive other investigational therapy, if available. The study doctor will discuss the possible risks and benefits of these treatments. You may choose not to have treatment for cancer at all. In all cases, you will receive appropriate medical care, including treatment for pain and other symptoms of cancer.

#### 1. STUDY DETAILS

## **Screening Tests**

Signing this consent form does not mean that you will be able to take part in this study. The following screening tests will help the doctor decide if you are eligible:

- You will have a physical exam.
- You will have an EKG to check your heart function.
- Blood (about 2½ tablespoons) will be drawn for routine tests, for biomarker testing, and to test for viruses (like hepatitis B and C and HIV [the AIDS virus]). Biomarkers are found in the blood/tissue and may be related to your reaction to the study drugs.
- Urine will be collected for routine tests.
- You will have a CT or PET/CT scan to check the status of the disease.
- If available, leftover tumor tissue from a previous procedure will be collected to confirm your diagnosis and to be used for biomarker testing. If not available, you will have a tumor biopsy. The study doctor will tell what type of biopsy you will have and explain its risks.
- If you can become pregnant, part of the above blood or urine sample will be used for a pregnancy test. To take part in this study, you must not be pregnant.

The study doctor will discuss the screening test results with you. If the screening tests show that you are not eligible to take part in the study, you will not be enrolled. Other treatment options will be discussed with you.

Up to 16 participants will be enrolled in this study. All will take part at MD Anderson.

# **Study Drug Administration**

Each study cycle is 21 days (3 weeks).

You will receive pembrolizumab by vein over about 30 minutes every 3 weeks during Weeks 1-10.

Every 2 weeks for 8 weeks, you will receive mFOLFOX6:

- Oxaliplatin by vein over about 2 hours
- 5-FU by vein non-stop (continuously) for 48 hours (over about 2 days)

During Weeks 9-13, you will not receive any treatment.

Then, during Weeks 13-18:

- You will receive 5-FU by vein non-stop for 5 days in a row (for example, Monday through Friday) each week.
- You will receive docetaxel by vein over about 1 hour 1 time every week.
- You will receive radiation therapy. You will sign a separate informed consent document that explains how and when you will receive radiation therapy, including its risks.

After Week 18, you will not receive any treatment for about 6-9 weeks.

Starting at either Week 24 or Week 27 (depending on when your doctor thinks you should begin receiving the study drug again), you will receive pembrolizumab again. You will continue to receive pembrolizumab every 6 weeks until Cycle 20 or until the disease gets worse.

You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

## **Study Visits**

#### On Day 1 of all cycles:

- You will have a physical exam.
- Blood (about 1½-2 tablespoons) will be drawn for routine tests. During Cycles 3 and 6, this blood will also be used for biomarker testing.
- You will have a tumor biopsy for biomarker testing during Cycles 3 and 6.
- If you can become pregnant, urine will be collected for a pregnancy test.

Once a week during Weeks 13-18, you will be asked how you are doing by the study staff. This will be done during a remote visit or in person.

**Every 9 weeks until Week 54 and then every 12 weeks after that**, you will have a CT or PET/CT scan to check the status of the disease.

# **End-of-Treatment Visit**

As soon as possible after your last dose of pembrolizumab:

- You will have a physical exam.
- Blood (about 1½ tablespoons) will be drawn for routine tests.
- You will have a CT or PET/CT scan to check the status of the disease.

# Follow-Up

About 30 days after your last dose of study drugs:

- Blood (about 1 tablespoon) will be drawn for routine tests.
- If you can become pregnant, blood (about 1 tablespoon) or urine will be collected for a pregnancy test.

# **Long-Term Follow-Up**

After your 30-day follow-up visit, if you stopped taking the study drugs for reasons other than the disease getting worse, you will continue to come to the clinic every 9-12 weeks to have a CT or PET/CT scan. If you start a new anti-cancer therapy or the disease gets worse, you will stop having imaging scans.

If you stopped taking the study drugs because the disease got worse or you started a new anti-cancer therapy, you will be called by the study staff about every 12 weeks until you withdraw from the study/the study ends.

#### 2. POSSIBLE RISKS

While on this study, you are at risk for side effects. You should discuss these with the study doctor. The more commonly occurring side effects are listed in this form, as are rare but serious side effects. You may also want to ask about uncommon side effects that have been observed in small numbers of patients but are not listed in this form. Many side effects go away shortly after treatment is stopped, but in some cases side effects may be serious, long-lasting or permanent, and may even result in hospitalization and/or death.

Side effects will vary from person to person, and some may occur after you have stopped receiving treatment. Tell the study staff about any side effects you may have, even if you do not think they are related to the study drugs/procedures.

## **Pembrolizumab Side Effects**

Common (occurring in more than 20% of patients)

- fatigue
- fever
- skin rash and/or itching
- abnormal salts,
  minerals, and/or acids
  in the blood (possible
  weakness, swelling,
  fatigue, low blood
  pressure, organ failure,
  heart problems,
  changes in mental
  status, and/or seizure)
- high blood sugar (possible diabetes)
- high blood levels of fat (possible heart disease and/or stroke)
- loss of appetite
- nausea
- constipation
- diarrhea
- abdominal pain
- low blood cell count (white/red/platelets)

- abnormal liver test (possible liver damage)
- pain
- abnormal kidney test (possible kidney damage)
- cough
- · difficulty breathing

Pembrolizumab may commonly cause low blood cell counts (red blood cells, platelets, and white blood cells):

- A low red blood cell count (anemia) may cause difficulty breathing and/or fatigue. You may need a blood transfusion.
- A low platelet count increases your risk of bleeding (such as nosebleeds, bruising, stroke, and/or digestive system bleeding). You may need a platelet transfusion.
- A low white blood cell count increases your risk of infection (such as pneumonia and/or severe blood infection). Infections may occur anywhere and become lifethreatening. Symptoms of infection may include fever, pain, redness, and difficulty breathing.

# Occasional (occurring in 3-20% of patients)

- swelling (face/arm/leg)
- inflammation of the tissue around the heart (possible chest pain)
- irregular heartbeat
- headache
- confusion
- patches of skin color loss
- underactive thyroid gland (possible weight gain, heart failure, and/or constipation)
- overactive thyroid gland (possible weight loss, diarrhea, mood swings, difficulty sleeping, heart rate changes, and/or sweating)
- low blood sugar
- weight loss
- fluid in the abdomen
- blood in the urine
- vomiting
- abnormal liver test (possible yellowing of the skin and/or eyes)
- weakness

- nerve damage (possible numbness, pain, and/or loss of motor function)
- difficulty breathing (possibly due to lung inflammation)
- flu-like symptoms
- infusion reaction (possible dizziness, low blood pressure, nausea, pain, and/or difficulty breathing

# Frequency Unknown

- heart failure
- heart attack
- build-up of fluid around the heart (possible heart failure)
- abnormal connections or passageways between organs or vessels
- bleeding in the rectum and/or uterus
- blockage in the lung (possible pain and/or shortness of breath)
- nosebleed
- coughing up blood

# Rare but serious (occurring in fewer than 3% of patients)

- low blood pressure (possible dizziness/fainting)
- heart inflammation
- build-up of fluid in the tissue around the heart
- blood vessel inflammation (possible bleeding, skin rash, numbness/weakness, fever, weight loss, fatigue, and/or bruising, depending on where the inflammation occurs)
- seizure
- immune system damage to the nervous system (causing muscle weakness, numbness and/or paralysis)
- spinal cord inflammation (possible pain, weakness, loss of feeling or movement, and/or paralysis)
- brain inflammation (possible paralysis and/or coma)
- shedding, scaling and/or inflammation of the skin (possible

- low hormone blood levels (possible weakness, bone changes, and/or cramping)
- hormonal deficiency that affects the body's ability to control blood pressure and react to stress
- pituitary gland inflammation (possible headaches)
- inflammation of the thyroid gland (possible tenderness in the neck)
- diabetes requiring insulin
- severe high blood sugar due to uncontrolled diabetes
- decreased production of adrenal hormones (possible weakness and/or low blood pressure)
- low pancreatic enzyme level (possible bloating, gas, abdominal discomfort, diarrhea, oily stool, and/or weight loss)

- inflammation inside the eye (possible vision problems)
- kidney inflammation (possible kidney damage/failure)
- kidney failure
- inflammation of an eye nerve (possible vision loss, loss of color vision, pain when moving your eyes, and/or loss of peripheral vision in one or both eyes)
- build-up of fluid around the lungs
- immune response that causes the body to attack itself (possible organ damage)
- multi-organ disease causing lesions, most often in the lungs (sarcoidosis)
- immune response (causing muscle weakness)
- immune system reaction (possible fever, jaundice, liver/spleen enlargement, irritability, and/or seizures)

- fatal loss of bodily fluids)
- large skin blisters
- very severe blistering skin disease (loss of large portion of skin and/or with ulcers of the skin and digestive tract)
- inflammation of the pancreas (possible abdominal pain)
- inflammation of the stomach (possible belly pain, fullness, nausea, vomiting, and/or loss of appetite)
- inflammation of the intestines (possibly with a hole in the intestines, which may lead to contents leaking into the abdomen)
- anemia due to destruction of red blood cells
- liver damage (hepatitis)
- inflammation/scarring of the bile ducts (tubes that carry digestive fluid that is made in the liver) liver damage, stomach pain, yellowing of the skin/eyes, fatigue, and/or itching)

- severe lifethreatening infection (possible low blood pressure, kidney failure, and/or heart failure)
- Vogt Koyanagi
   Harada syndrome pigmented tissue
   (possible eye
   pain/swelling and
   changes in vision,
   hearing loss, and/or
   white patches on the
   skin)
- low number of red blood cells (cells that carry oxygen) due to destruction of red blood cells (hemolytic anemia). You may feel weak, tired, lightheaded, short of breath, or have a fast heartbeat. You may also experience difficulty with physical exercise, pale or yellow skin, dark urine, or fever
- Inflammation of the protective sac surrounding your heart (pericarditis) which can cause sharp chest pain and shortness of breath (especially when lying flat), fever, and a fast or irregular heartbeat. In severe cases, your heart may have difficulty

| pumping blood |
|-----------------|
| throughout your |
| body. |

If you have a solid tumor type and you have an organ transplant, pembrolizumab may increase your risk for the transplant to be rejected by your body.

Pembrolizumab works by boosting the immune system. This may cause unknown side effects resulting from your immune system attacking your organs. This may cause inflammation and inflammation-related side effects in any organ or tissue. These side effects can affect more than one of your normal organs and tissues at the same time.

If you have a stem cell transplant from a donor after you receive pembrolizumab, you may have an increased risk of complications, such as severe graft-versus-host disease (when transplanted donor tissue attacks the recipient's organs such as skin, liver, and/or intestines) and/or clotting of blood within the liver. Deaths have been reported in patients who received a stem cell transplant from a donor after pembrolizumab therapy. If you decide to receive a stem cell transplant from a donor, please tell your transplant doctor that you received pembrolizumab in the past.

# Side Effects for Oxaliplatin, 5-FU, and Docetaxel

Only pembrolizumab is supplied by the study sponsor. The other drugs (oxaliplatin, 5-FU, and docetaxel) are considered part of standard care for the disease. You will be given a second consent document to sign that contains current information on the risks and side effects related to those drugs. You will have a chance to ask the study team any questions you have about those drugs and their side effects. You will also be informed of any important new information about those drugs that may affect your willingness to continue taking part in this study.

**Using the study drugs together** may cause side effects that are not seen when each drug is given alone. The study drug combination may also increase the frequency and/or severity of the side effects listed above.

#### Other Risks

**Blood draws** may cause pain, bleeding, and/or bruising. You may faint and/or develop an infection with redness and irritation of the vein at the site where blood is drawn. Frequent blood collection may cause anemia (low red blood cell count), which may create a need for blood transfusions.

**EKGs** may cause discomfort while lying on the exam table, and the tape on the EKG pads may cause skin irritation.

A **PET scan** may cause you to feel "closed in" while lying in the scanner. However, the scanner is open at both ends and an intercom allows you to talk with doctors and staff. If you feel ill or anxious during scanning, doctors and/or technicians will give comfort or the scanning will be stopped.

The PET scan exposes your body to radiation. The radioactive solution does not remain in your system for a long period of time. However, you should wait 2 hours before holding an infant or getting close to a pregnant woman to avoid exposing them to radiation. You should drink fluids after the scan to help remove the solution from your system.

CT scans send x-rays through the body at many different angles. You will be exposed to a small dose of radiation. All radiation adds up over a lifetime and may increase the risk of new cancer forming. Some people may feel "closed in" while lying in the scanner. However, the scanner is open at both ends, and an intercom allows you to talk with doctors and staff. If you feel ill or anxious during scanning, doctors and/or radiology technicians will give comfort, or the scanning will be stopped. When a CT scan of the abdominal area is taken, material may be inserted into the rectum to better define the bowel. You will usually drink liquid to help define various abdominal organs. This may cause nausea and/or vomiting. Solution may also be given by vein to make the x-ray pictures more accurate. This may cause an uncomfortable feeling of warmth, nausea, and/or severe allergic reactions. The solution injection may also cause pain, bleeding, bruising, hives, and/or itching.

Having **biopsies** performed may cause pain, bruising, bleeding, redness, low blood pressure, swelling, and/or infection at the site of the biopsies. An allergic reaction to the anesthetic may occur. A scar may form at the biopsy site.

Although every effort will be made to keep study data safe, there is a chance that your personal health information could be lost or stolen, which may result in a **loss of confidentiality**. All study data will be stored in password-protected computers and/or locked file cabinets and will continue to be stored securely after the study.

This study may involve unpredictable risks to the participants.

# **Pregnancy Related Risks**

Taking part in this study can result in risks to an unborn or breastfeeding baby, so you should not become pregnant, breastfeed a baby, or father a child while on this study. You must use birth control during the study if you are sexually active.

Birth Control Specifications: If you can become pregnant or father a child, you must use a highly effective method of birth control during the study and for 180 days after taking the study drugs. Acceptable methods of birth control include:

- Combined (estrogen- and progestogen-containing) hormonal birth control (including pills, patches, or injections)
- Progestogen-only hormonal birth control (pills, injections, or implants)
- Intrauterine hormone-releasing system (IUS) or device (IUD)
- Bilateral tubal occlusion ("tubes tied")
- Vasectomy of yourself or a partner

Males: Do not donate sperm while on this study. Tell the doctor right away if your partner becomes pregnant or suspects pregnancy.

Females: If you are pregnant, you will not be enrolled on this study. If you become pregnant or suspect that you are pregnant, you must tell your doctor right away.

Getting pregnant will result in your removal from this study.

## **OPTIONAL PROCEDURES FOR THE STUDY**

**Optional Procedure #1:** If you agree, blood (1 teaspoon) will be drawn for biomarker testing at the end-of-treatment visit.

**Optional Procedure #2:** If you agree, you will have a tumor biopsy for biomarker testing at the end-of-treatment visit.

There are no benefits to you for taking part in the optional procedures. Future patients may benefit from what is learned. You may stop taking part at any time. There will be no cost to you for taking part in the optional procedures.

# **Optional Procedure Risks**

**Blood draws** may cause pain, bleeding, and/or bruising. You may faint and/or develop an infection with redness and irritation of the vein at the site where blood is drawn. Frequent blood collection may cause anemia (low red blood cell count), which may create a need for blood transfusions.

Having **biopsies** performed may cause pain, bruising, bleeding, redness, low blood pressure, swelling, and/or infection at the site of the biopsies. An allergic reaction to the anesthetic may occur. A scar may form at the biopsy site.

#### CONSENT/PERMISSION/AUTHORIZATION FOR OPTIONAL PROCEDURES

Circle your choice of "yes" or "no" for each of the following optional procedures:

**Optional Procedure #1:** Do you agree to have additional blood drawn for biomarker testing?

YES NO

Optional Procedure #2: Do you agree to have a tumor biopsy for biomarker testing?

YES NO

#### 3. COSTS AND COMPENSATION

If you suffer injury as a direct result of taking part in this study, MD Anderson health providers will provide medical care. However, this medical care will be billed to your insurance provider or you in the ordinary manner. You will not be reimbursed for expenses or compensated financially by MD Anderson for this injury. You may also contact the Chair of MD Anderson's IRB at 713-792-6477 with questions about study-related injuries. By signing this consent form, you are not giving up any of your legal rights.

If you become injured or ill as a direct result of taking part in this study, the sponsor may pay for the treatment of the injury or illness. MD Anderson cannot determine at this time what you may be reimbursed for. A financial counselor will be made available to you after the injury or illness is reported.

Certain tests, procedures, and/or drugs that you may receive as part of this study may be without cost to you because they are for research purposes only. However, your insurance provider and/or you may be financially responsible for the cost of care and treatment of any complications resulting from the research tests, procedures, and/or drugs. Standard medical care that you receive under this research study will be billed to your insurance provider and/or you in the ordinary manner. Before taking part in this study, you may ask about which parts of the research-related care may be provided without charge, which costs your insurance provider may pay for, and which costs may be your responsibility. You may ask that a financial counselor be made available to you to talk about the costs of this study.

Samples that are collected from you in this study may be used for the development of treatments, devices, new drugs, or patentable procedures that may result in commercial profit.

There are no plans to compensate you for any patents or discoveries that may result from your participation in this research.

You will receive no compensation for taking part in this study.

## **Additional Information**

- 4. You may ask the study chair (Dr. Jaffer Ajani, at 713-792-2828) any questions you have about this study. You may also contact the Chair of MD Anderson's Institutional Review Board (IRB a committee that reviews research studies) at 713-792-6477 with any questions that have to do with this study or your rights as a study participant.
- 5. You may choose not to take part in this study without any penalty or loss of benefits to which you are otherwise entitled. You may also withdraw from participation in this study at any time without any penalty or loss of benefits. If you decide you want to stop taking part in the study, it is recommended for your safety that you first talk to your doctor. It may be dangerous to suddenly stop study treatment, so you may be asked to come back to the clinic for more safety tests or other procedures. If you withdraw from this study, you can still choose to

be treated at MD Anderson.

If you stop being in the research, already collected data may not be removed from the study database. You may be asked whether the study doctor can collect data from your routine medical care. If you agree, this data will be handled the same as research data.

- 6. This study or your participation in it may be changed or stopped without your consent at any time by the study chair, Merck, the U.S. Food and Drug Administration (FDA), the Office for Human Research Protections (OHRP), or the IRB of MD Anderson.
- 7. You will be informed of any new findings or information that might affect your willingness to continue taking part in the study, including the results of all of your standard tests performed as part of this research, and you may be asked to sign another informed consent and authorization form stating your continued willingness to participate in this study.

The results of any genetic tests will not be put in your health records.

- 8. MD Anderson may benefit from your participation and/or what is learned in this study.
- 9. This study is sponsored and/or supported by: Merck.
- 10. In a medical emergency, you may be cared for by someone who has a financial interest with the study sponsor(s)/supporter. If you have any questions about this, you may call the IRB at 713-792-6477.

## **Future Research**

#### Data

Your personal information is being collected as part of this study. These data may be used by researchers at MD Anderson and Merck and/or shared with other researchers and/or institutions for use in future research.

If you do not want your samples or data to be used for future research, tell the study doctor. You may withdraw your samples at any time by telling your study team. If you decide to withdraw your samples, they will be returned to the lab they came from or destroyed. However, the data and test results already collected from your samples will be kept and may be used.

#### Samples

Samples (such as blood and/or tissue) are being collected from you as part of this study. Researchers at MD Anderson may use any leftover samples that are stored at MD Anderson in future research. Leftover samples stored by Merck may be used in future research. Your samples will be stored for up to 15 years after the study ends. After this time, they will be destroyed.

Before being used or shared for future research, every effort will be made to remove your identifying information from any data and/or research samples. If all identifying information is removed, you will not be asked for additional permission before future research is performed.

In some cases, all of your identifying information may not be removed before your data or research samples are used for future research. If future research is performed at MD Anderson, the researchers must get approval from the Institutional Review Board (IRB) of MD Anderson before your data and/or research samples can be used. At that time, the IRB will decide whether or not further permission from you is required. The IRB is a committee of doctors, researchers, and community members that is responsible for protecting study participants and making sure all research is safe and ethical.

If this research is not performed at MD Anderson, MD Anderson will not have oversight of any data and/or samples.

#### **Genetic Research**

Research samples collected from you as part of this study may be used for genetic research, which may include whole genome sequencing. Whole genome sequencing is a type of testing in which researchers study your entire genetic makeup (DNA). This may help researchers learn how changes in the ordering of genes may affect a disease or response to treatment.

A federal law, called the Genetic Information Nondiscrimination Act (GINA), generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. This law generally will protect you in the following ways:

- Health insurance companies and group health plans may not request your genetic information that we get from this research.
- Health insurance companies and group health plans may not use your genetic information when making decisions regarding your eligibility or premiums.
- Employers with 15 or more employees may not use your genetic information that we get from this research when deciding to hire, promote, or fire you or when setting the terms of your employment.

Be aware that this federal law does not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. Nor does this federal law prohibit discrimination based on an already known genetic disease or disorder.

#### **Conflict of Interest**

Outside relationships are disclosed to and approved by the Conflict of Interest Committee, which reviews these relationships for compliance with institutional policy. This review helps the IRB to assure that financial relationships do not have an impact on the conduct of this study. The following members of the study staff have disclosed compensation from the funding source(s) of this study:

Dr. Jaffer Ajani (Study Chair)

# <u>Authorization for Use and Disclosure of Protected Health Information (PHI):</u>

- A. During the course of this study, MD Anderson will be collecting and using your PHI, including identifying information, information from your medical record, and study results. For legal, ethical, research, and safety-related reasons, your doctor and the research team may share your PHI with:
  - Federal agencies that require reporting of clinical study data (such as the FDA, National Cancer Institute [NCI], and OHRP)
  - The IRB and officials of MD Anderson
  - Other companies in the AstraZeneca group, service providers, contractors, and research institutions that support this study
  - ICON Clinical Research
  - Study monitors and auditors who verify the accuracy of the information
  - Individuals who put all the study information together in report form

Merck may receive limited amounts of PHI as a research partner. They may also view additional PHI in study records during the monitoring process. MD Anderson's contracts require research partners to protect this information and limit how they may use it.

As part of their oversight, the FDA also review your study records.

To protect your identity, the samples collected from you will be labeled a unique number instead of your name or other identifying information. Only the study doctor or study staff will have access to the code that can link you to your samples.

If results from this study are published, such as in medical journals or online, your name and other identifying information will not be used.

- B. Signing this consent and authorization form is optional but you cannot take part in this study or receive study-related treatment if you do not agree and sign.
- C. MD Anderson will do its best to protect the privacy of your records, but it is possible that once information is shared with people listed on this form, it may be released to others. If this happens, your information may no longer be protected by federal law.

- D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected.
- E. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# **CONSENT/AUTHORIZATION**

I understand the information in this consent form. I have had a chance to read the

consent form for this study, or have had it read to me. I have had a chance to think about it, ask questions, and talk about it with others as needed. I give the study chair permission to enroll me on this study. By signing this consent form, I am not giving up any of my legal rights. I will be given a signed copy of this consent document. SIGNATURE OF PARTICIPANT DATE PRINTED NAME OF PARTICIPANT **WITNESS TO CONSENT** I was present during the explanation of the research to be performed under this protocol. SIGNATURE OF WITNESS TO THE VERBAL CONSENT DATE PRESENTATION (OTHER THAN PHYSICIAN OR STUDY CHAIR) A witness signature is only required for non-English speakers utilizing the short form consent process (VTPS) and patients who are illiterate. PRINTED NAME OF WITNESS TO THE VERBAL CONSENT PERSON OBTAINING CONSENT I have discussed this research study with the participant and/or his or her authorized representative, using language that is understandable and appropriate. I believe that I have fully informed this participant of the nature of this study and its possible benefits and risks and that the participant understood this explanation. PERSON OBTAINING CONSENT DATE PRINTED NAME OF PERSON OBTAINING CONSENT